CLINICAL TRIAL: NCT02925949
Title: A Couples-based Approach to Improving Engagement in HIV Care
Brief Title: Duo Partnership Adherence Commitment Therapy
Acronym: DuoPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2R01NR010187-10A1 (NIH); 2R01NR010187-10A1 (NIH)
Record Dates: First submitted 2016-09-28; First posted 2016-10-06 (Estimated); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: HIV/AIDS
Keywords: Treatment; Adherence; Intervention; Sexual and Gender Minority Couples
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Coitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DuoPACT (Active Comparator): A 6-session HIV medication adherence support program for couples.
  Interventions: Behavioral: DuoPACT
- LifeSteps (Active Comparator): A 3-session HIV medication adherence support program for individuals.
  Interventions: Behavioral: LifeSteps

INTERVENTIONS:
Behavioral: DuoPACT — 6 couple-based intervention sessions are administered weekly by a counselor.
  Arms: DuoPACT
Behavioral: LifeSteps — 3 individual-based intervention sessions are administered weekly by a counselor.
  Arms: LifeSteps

SUMMARY:
This is a randomized controlled trial of a new behavioral intervention designed to improve engagement in HIV care for couples. Investigators will compare the HIV viral load outcomes of couples randomized to a couples-based adherence intervention (DuoPACT) or to an individual adherence intervention (LifeSteps).

DETAILED DESCRIPTION:
The investigators will test the intervention to improve HIV care engagement by enrolling 150 sexual or gender minority couples and randomizing 75 couples each to one of two conditions: 1) DuoPACT, a newly-developed couples intervention; or 2) LifeSteps, a standardized antiretroviral adherence intervention for HIV+ individuals. After randomization, intervention sessions will be delivered weekly (6 DuoPACT sessions, or 3 Life Steps sessions). All couples will be assessed pre/post intervention to evaluate intervention effects via behavioral indicators of engagement in HIV care, the couple's relationship dynamics, and the primary outcome of HIV viral load.

ELIGIBILITY:
Inclusion Criteria:

1. 18+ years old;
2. Identifies as a sexual or gender minority;
3. In a primary romantic relationship for at least 3 months;
4. At least one partner is HIV+;
5. English-speaking;
6. Able to provide informed consent; and
7. For HIV+ participants: Evidence of suboptimal engagement in HIV care.

Exclusion Criteria:

1. Must be able to consent to and follow study protocol;
2. Evidence of severe cognitive impairment or active psychosis;
3. Lives outside California or plans to relocate from the state of California in the next 6 months; or
4. Participation in the DuoPACT pilot.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Sexual and Gender Minorities
Enrollment: 288 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline HIV viral load at 3, 6 and 9 months | 3, 6 and 9 months
  Follow-up blood draws will be performed on all HIV+ partners at 3, 6, and 9 months post randomization. HIV-1 viral load levels will be measured by the COBAS® AmpliPrep/COBAS® TaqMan® HIV test kit (Roche Molecular Systems, Inc.), which has a threshold for undetectability = < 20 copies/mL.

SECONDARY OUTCOMES:
Change from Baseline behavioral indicators of engagement in HIV care at 3, 6 and 9 months | 3, 6 and 9 months
  The investigators will use a newly developed 8-point scale called the Behavioral Composite of Engagement in HIV Care, which integrates:
  * Current/past ART use (participant self-report and verification by HIV medication pill bottles or current pharmacy prescription).
  * HIV appointment attendance (participant self-report categorized according to current HRSA standards of the minimum annual number and spacing of HIV primary care appointments).
  * ART adherence (participant self-report and Walsh visual analog scale),
  * Knowledge of current CD4 cell count (participant self-report).

CONTACTS AND LOCATIONS:
Overall Officials: Mallory O. Johnson, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Center for AIDS Prevention Studies, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
A de-identified dataset will be made available to investigators upon reasonable request and following completion of primary study analyses.

REFERENCES:
- [Background] Tabrisky AP, Coffin LS, Olem DP, Neilands TB, Johnson MO. Couples-focused intervention to improve engagement in HIV care: protocol for a randomised controlled trial. BMJ Open. 2021 Mar 22;11(3):e037468. doi: 10.1136/bmjopen-2020-037468. PMID 33753428
- See also: Couples-focused intervention to improve engagement in HIV care: protocol for a randomised controlled trial — https://pubmed.ncbi.nlm.nih.gov/33753428/